CLINICAL TRIAL: NCT07252401
Title: Terlipressin vs. Somatostatin in Cirrhotic Patients With Acute Gastrointestinal Bleeding and Acute Kidney Injury: A Multicenter Randomized Controlled Trial
Brief Title: Terlipressin vs. Somatostatin in Cirrhotic Patients With Acute Gastrointestinal Bleeding and Acute Kidney Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Director of Department of Gastroenterology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TERLI-AGIB-AKI
Record Dates: First submitted 2025-11-16; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Liver Cirrhosis
Keywords: acute gastrointestinal bleeding; acute kidney injury; terlipressin; somatostatin; liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Acute Kidney Injury | interventions — Terlipressin; terlivaz; Somatostatin

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Terlipressin group (Experimental): Continuous intravenous infusion of terlipressin 2-4 mg every 12 hours.
  Interventions: Drug: 2-4 mg of terlipressin
- Somatostatin group (Active Comparator): Continuous intravenous infusion of somatostatin 3 mg every 12 hours.
  Interventions: Drug: 3 mg of somatostatin

INTERVENTIONS:
Drug: 2-4 mg of terlipressin — Participants receive 2-4 mg of terlipressin by continuous intravenous infusion every 12 hours, with a maximum treatment course of 5 days.
  Other Names: Terlivaz
  Arms: Terlipressin group
Drug: 3 mg of somatostatin — Participants receive 3 mg of somatostatin by continuous intravenous infusion every 12 hours, with a maximum treatment course of 5 days.
  Other Names: Stilamin
  Arms: Somatostatin group

SUMMARY:
Acute gastrointestinal bleeding (AGIB) is a common complication in the decompensated stage of liver cirrhosis, of which approximately 70% is acute variceal bleeding (AVB) caused by portal hypertension. Existing evidence suggests that both terlipressin and somatostatin can be used to control AVB in cirrhotic patients, but terlipressin may be the first-line treatment for cirrhotic patients with AGIB complicated by acute kidney injury (AKI). Herein, a multicenter randomized controlled trial (RCT) has been designed to compare the efficacy of terlipressin and somatostatin in the treatment of cirrhotic patients with AGIB complicated by AKI.

DETAILED DESCRIPTION:
Overall, 64 cirrhotic patients with a diagnosis of AGIB and AKI will be enrolled. They will be stratified according to the severity of AKI, and then randomly assigned to terlipressin group and somatostatin group at a ratio of 1:1. The primary endpoint is reversal of AKI after treatment on 5 days. Secondary endpoints include duration of AKI, recurrence of AKI, rates of renal replacement therapy, transjugular intrahepatic portosystemic shunt (TIPS) treatment, liver, and kidney transplantation, 6-week mortality, 6-week rebleeding rate, and incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* patients have a definite diagnosis of live cirrhosis and AKI;
* patients present with AGIB at admission;
* patients' age 18-70 years old;
* patients or relatives can sign the informed consent form.

Exclusion Criteria:

* patients have hepatorenal syndrome- acute renal injury (HRS-AKI);
* patients have structural kidney injury;
* patients have chronic kidney disease;
* patients received terlipressin or somatostatin therapy within 48 hours before enrollment;
* patients received kidney replacement therapy before enrollment;
* patients have a history of liver transplantation or TIPS;
* patients have acute liver failure or acute-on-chronic liver failure;
* patients have hepatic or renal malignant tumor;
* patients have severe diseases of the heart, lungs, and brain;
* patients have contraindications for experimental drugs;
* patients are in pregnancy or lactation;
* patients participated in other clinical studies within 3 months before enrollment;
* patients have other conditions that investigators deem unsuitable for enrollment in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Reversal of AKI | 5 days
  The reversal of AKI is defined as clinical symptoms of AKI disappear and serum creatinine (SCr) levels decrease after treatment.

SECONDARY OUTCOMES:
Duration of AKI | 6 weeks
  The duration of AKI is defined as the time from occurrence to reversal of AKI.
Recurrence of AKI | 6 weeks
  Clinical symptoms related to AKI recur and SCr levels increase after the reserval of AKI. The diagnosis of AKI should meet any of the following conditions: an increase in SCr level of ≥0.3 mg/dl (26.5 μmol/L) within 48 hours; or an increase in SCr level to ≥1.5 times the baseline value within 7 days; or urine output <0.5 ml/kg per hour for a continuous 6 hours.
Kidney replacement therapy rate | 6 weeks
  Participants undergo dialysis or continuous kidney replacement therapy due to failure to recover renal function after treatment.
Transjugular intrahepatic portosystemic shunt (TIPS) treatment rate | 6 weeks
  Participants undergo transjugular intrahepatic portosystemic shunt (TIPS) treatment.
Liver and kidney transplantation treatment rate | 6 weeks
  Participants undergo liver and kidney transplantation treatment.
6-week mortality rate | 6 weeks
  The 6-week mortality rate is defined as the all-cause mortality rate over 6 weeks.
6-week rebleeding rate | 6 weeks
  The 6-week rebleeding rate is defined as the rebleeding rate within 6 weeks after successful AVB hemostasis.
Adverse events | 6 weeks
  Adverse events will be monitored, including nausea, abdominal pain, diarrhea, arrhythmia, dyspnea, and hyponatremia that may be caused by terlipressin, as well as nausea, abdominal pain, diarrhea, hypoglycemia, and allergies that may be caused by somatostatin.

CONTACTS AND LOCATIONS:
Overall Officials: Xingshun Qi, MD, Principal Investigator — Department of Gastroenterology, General Hospital of Northern Theater Command; Qianqian Li, Principal Investigator — Department of Gastroenterology, General Hospital of Northern Theater Command; Rong Li, Principal Investigator — Department of Gastroenterology, General Hospital of Northern Theater Command
Locations (1):
- Department of Gastroenterology, General Hospital of Northern Theater Command (formerly called General Hospital of Shenyang Military Area), Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Xu X, Liu B, Lin S, Li B, Wu Y, Li Y, Zhu Q, Yang Y, Tang S, Meng F, Chen Y, Yuan S, Shao L, Bernardi M, Yoshida EM, Qi X. Terlipressin May Decrease In-Hospital Mortality of Cirrhotic Patients with Acute Gastrointestinal Bleeding and Renal Dysfunction: A Retrospective Multicenter Observational Study. Adv Ther. 2020 Oct;37(10):4396-4413. doi: 10.1007/s12325-020-01466-z. Epub 2020 Aug 28. PMID 32860184
- [Result] Walker S, Kreichgauer HP, Bode JC. Terlipressin vs. somatostatin in bleeding esophageal varices: a controlled, double-blind study. Hepatology. 1992 Jun;15(6):1023-30. doi: 10.1002/hep.1840150609. PMID 1350562
- [Result] Zhou X, Tripathi D, Song T, Shao L, Han B, Zhu J, Han D, Liu F, Qi X. Terlipressin for the treatment of acute variceal bleeding: A systematic review and meta-analysis of randomized controlled trials. Medicine (Baltimore). 2018 Nov;97(48):e13437. doi: 10.1097/MD.0000000000013437. PMID 30508958
- [Result] Xu X, Tang C, Linghu E, Ding H; Chinese Society of Hepatology, Chinese Medical Association; Chinese Society of Gastroenterology, Chinese Medical Association; Chinese Society of Digestive Endoscopy, Chinese Medical Association. Guidelines for the Management of Esophagogastric Variceal Bleeding in Cirrhotic Portal Hypertension. J Clin Transl Hepatol. 2023 Dec 28;11(7):1565-1579. doi: 10.14218/JCTH.2023.00061. Epub 2023 Oct 17. PMID 38161497